CLINICAL TRIAL: NCT00452062
Title: Mackay Memorial Hospital
Brief Title: Dexamethasone and the Prevention of Post-Extubation Airway Obstruction in Adults
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mackay Memorial Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: MMH-I-S-106
Record Dates: First submitted 2007-03-23; First posted 2007-03-26 (Estimated); Last update posted 2007-03-26 (Estimated); Status verified 2007-03

CONDITIONS: Airway Obstruction
Keywords: cuff-leak test; intubation; corticosteroids; dexamethasone to reduce the occurrence of post-extubation airway obstruction
MeSH Terms: conditions — Airway Obstruction | interventions — Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Dexamethasone

SUMMARY:
Laryngotracheal injury related to intubation may cause narrowing of the airway due to edema of the glottis. Post-extubation airway frequently necessitating re-intubation and resulting in the prolongation of intensive care. Factors correlating with the development of post-extubation stridor include age, female gender, an elevated Acute Physiologic and Chronic Health Evaluation II, trauma related to endotracheal intubation, excessive ETT size, unnecessary tube mobility, increased cuff pressure, frequent tracheal aspirations, infection, arterial hypotension, and a prolonged intubation period. Because the presence of an endotracheal tube (ETT) precludes direct visualization of the upper airway, recognition of edema due to laryngotracheal injury is often difficult. However, upper airway patency may be measured indirectly in the intubated patient by documentation of a leak around the ETT upon deflation of the sealing balloon cuff encircling the ETT. Controversy currently exists regarding the effectiveness of prophylactic steroid therapy for patients considered at high risk for post-extubation stridor. Only a limited number of prospective trials involving adults and evaluating the benefits of corticosteroid therapy prior to extubation have been conducted.

Studies regarding the efficacy of prophylactic corticosteroids for intubated patients have yielded conflicting results due to differences in the number of doses or types of corticosteroids administered.

The present study was conducted to evaluate the effects of prophylactic dexamethasone therapy for a subset of high-risk patients who had been intubated for > 48 hours and who were undergoing their first elective extubation in an ICU setting. The specific objectives were to determine whether multiple doses of dexamethasone are effective in the reduction or prevention of post-extubation airway obstruction in patients with a cuff leak volume (CLV) < 110 mL and to ascertain whether an aftereffect follows the discontinuation of dexamethasone.

DETAILED DESCRIPTION:
Materials and methods Patients The current study included patients admitted to the adult medical ICU of the Mackay Memorial Medical Center from 1 October 2004 and 1 July 2007 and who met the inclusion criteria described below. Informed consent was obtained from the patients or their relatives prior to entering the trial. This study was approved by the Institutional Research Ethics Board. The cuff-leak test was therefore administered to patients requiring mechanical ventilation for more than 48 hours. All patients were > 18 years of age and met the following weaning criteria: 1) temperature ≤ 38°C for > 8 hours, 2) discontinuous use of sedatives, 3) heart rate ≥ 70 and ≤ 130 /min, 4) systolic blood pressure (SBP) ≥ 80 mm Hg in the absence of vasopressors, 5) fraction of inspired oxygen (FiO2) ≤ 0.6, PaO2 ≥ 60, and partial pressure of oxygen (PaO2)/FiO2 ratio > 200, 6) positive end-expiratory pressure (PEEP) ≤ 5 cm H2O, 7) rapid and shallow ratio of frequency to tidal volume (f/VT ≤ 105), 8) minute ventilation ≤ 15 L/min, and 9) pH ≥ 7.3. Supplemental oxygen was continued to maintain an oxygen saturation > 95% as measured by a pulse oximeter.

Exclusion criteria were: 1) the need for more than one tracheal intubation during the hospital stay, 2) unstable hemodynamics (i.e., a mean SBP < 90 mm Hg, a SBP decrease > 40 mm Hg, or a mean arterial pressure [MAP] < 70 mm Hg), 3) profound recalcitrant hypoxemia (i.e., PaO2 < 60 mm Hg with a FiO2 > 0.50), or 4) administration of corticosteroids 7 days prior to extubation. All patients were intubated with a high-volume, low-pressure cuffed ETT. Patients exhibiting excessive movement were sedated or paralyzed during mechanical ventilation. Routine nursing care included ETT suctioning every 2 hours or as needed to maintain a patent airway. Patients were mechanically ventilated in the volume-assisted control mode with a tidal volume of 10 mL/kg of ideal body weight, a respiratory rate of 20 breaths/minute, and a zero PEEP during CLV measurement. The operator-selected inspiratory tidal volume of 10 mL per kilogram of ideal body weight, displayed as an expiratory tidal volume, was recorded. The balloon cuff was deflated, the expiratory tidal volume was recorded over the 6 subsequent respiratory cycles, and the average of the lowest 3 values was utilized for subsequent analyses. The CLV was determined as the difference in the actual tidal volume before and after cuff deflation.

Study protocol Patients requiring mechanical ventilation for > 48 hours and exhibiting a CLV < 110 mL were therefore included in the trial. The study was prospective, randomized, double-blind, and placebo-controlled. The randomization procedure was performed by a respiratory therapist not involved in patient care using blocked randomization. Patients were randomized to receive intravenous dexamethasone 5 mg per injection, or intravenous normal saline at an equivalent volume. Dexamethasone or normal saline (placebo) was administered every 6 hours for a total of 4 doses. Cuff leak tests were measured one hour after each injection and 24 hours after the 4th injection of dexamethasone or placebo. Both the physician and the staff who administered the treatment were blinded. The ICU physicians were not apprised of the measurements obtained by the respiratory therapist. Extubation was carried out 24 hours after the last injection of intervention fluid. After extubation, the presence of an audible, high-pitched wheeze was an indication for the inhalation of racemic epinephrine.

Patients meeting at least two of the following criteria were assigned to take non-invasive positive-pressure ventilation by face mask: 1) respiratory acidosis (defined as an arterial pH < 7.35 with a partial pressure of arterial carbon dioxide > 45 mm Hg), 2) clinical signs suggestive of respiratory-muscle fatigue or increased respiratory effort (i.e., use of accessory muscles, intercostal retraction, or paradoxical motion of the abdomen), 3) a respiratory rate > 25 breaths per minute for 2 consecutive hours, and 4) hypoxemia (defined as an arterial oxygen saturation of < 90 % or a PaO2 of < 80 mm Hg with a FiO2 > 0.50). Patients were re-intubated with mechanical ventilation support if they met at least one of the following criteria: 1) pH < 7.3 with a partial pressure of carbon dioxide increase > 15 mm Hg, 2) a change in mental status rendering the patient unable to tolerate non-invasive ventilation, 3) a decrease in the oxygen saturation to < 85% despite the use of a high fraction of inspired oxygen (a PaO2 < 50 mm Hg with a FiO2 > 70 %), 4) lack of improvement in signs of respiratory-muscle fatigue, 5) hypotension with a SBP < 80 mm Hg for more than 30 minutes despite adequate volume challenge, 6) a diastolic blood pressure drop > 20 mm Hg, and 7) copious secretions that could not be adequately cleared or that were associated with acidosis, hypoxemia, or changes in mental status (somnolence, agitation, or diaphoresis).

ELIGIBILITY:
Inclusion Criteria:

All patients were > 18 years of age and met the following weaning criteria:

1. Temperature ≤ 38°C for > 8 hours,
2. Discontinuous use of sedatives,
3. Heart rate ≥ 70 and ≤ 130 /min,
4. Systolic blood pressure (SBP) ≥ 80 mm Hg in the absence of vasopressors,
5. Fraction of inspired oxygen (FiO2) ≤ 0.6, PaO2 ≥ 60, and partial pressure of oxygen (PaO2)/FiO2 ratio > 200,
6. Positive end-expiratory pressure (PEEP) ≤ 5 cm H2O,
7. Rapid and shallow ratio of frequency to tidal volume (f/VT ≤ 105),
8. Minute ventilation ≤ 15 L/min, and
9. pH ≥ 7.3. Supplemental oxygen was continued to maintain an oxygen saturation > 95% as measured by a pulse oximeter.

Exclusion Criteria:

1. The need for more than one tracheal intubation during the hospital stay,
2. Unstable hemodynamics (i.e., a mean SBP < 90 mm Hg, a SBP decrease > 40 mm Hg, or a mean arterial pressure [MAP] < 70 mm Hg),
3. Profound recalcitrant hypoxemia (i.e., PaO2 < 60 mm Hg with a FiO2 > 0.50), or
4. Administration of corticosteroids 7 days prior to extubation.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70
Dates: Start 2004-10; Study Completion 2007-07 (Estimated)

PRIMARY OUTCOMES:
The purpose of this study was to ascertain whether administration of multiple doses of dexamethasone to critically ill intubated patients reduces or prevents the occurrence of post-extubation airway obstruction.

SECONDARY OUTCOMES:
The secondary purpose of this study was to ascertain whether administration of multiple doses of dexamethasone to critically ill intubated patients reduces or prevents the occurrence of noninvasive ventilation or re-intubation.

CONTACTS AND LOCATIONS:
Overall Officials: Chao-Hsien Lee, MD, Principal Investigator — Mackay Memorial Hospital
Locations (1):
- Mackay Memorial Hospital, Taipei, Taipei, Taiwan

REFERENCES:
- [Result] Cheng KC, Hou CC, Huang HC, Lin SC, Zhang H. Intravenous injection of methylprednisolone reduces the incidence of postextubation stridor in intensive care unit patients. Crit Care Med. 2006 May;34(5):1345-50. doi: 10.1097/01.CCM.0000214678.92134.BD. PMID 16540947
- [Result] Anene O, Meert KL, Uy H, Simpson P, Sarnaik AP. Dexamethasone for the prevention of postextubation airway obstruction: a prospective, randomized, double-blind, placebo-controlled trial. Crit Care Med. 1996 Oct;24(10):1666-9. doi: 10.1097/00003246-199610000-00011. PMID 8874303
- [Result] Chung YH, Chao TY, Chiu CT, Lin MC. The cuff-leak test is a simple tool to verify severe laryngeal edema in patients undergoing long-term mechanical ventilation. Crit Care Med. 2006 Feb;34(2):409-14. doi: 10.1097/01.ccm.0000198105.65413.85. PMID 16424722
- [Derived] Lee CH, Peng MJ, Wu CL. Dexamethasone to prevent postextubation airway obstruction in adults: a prospective, randomized, double-blind, placebo-controlled study. Crit Care. 2007;11(4):R72. doi: 10.1186/cc5957. PMID 17605780